CLINICAL TRIAL: NCT03990012
Title: Infrared Imaging for Breast Cancer Modeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jody Hayes, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2018-0370
Record Dates: First submitted 2019-05-21; First posted 2019-06-18 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients referred for breast biopsy (Experimental): Patients with Breast Imaging-Reporting and Data System (BI-RADS) 4C or 5 diagnosis who have been referred for breast biopsy based on the results of their standard diagnostic breast exam will undergo IR and 3D imaging of the breasts.
  Interventions: Procedure: IR Imaging; Procedure: 3D Scanning

INTERVENTIONS:
Procedure: IR Imaging — Subjects will undergo steady steady state and video IR imaging of the breasts.
Procedure: 3D Scanning — Subjects will undergo 3D scanning of the breasts.

SUMMARY:
The primary objective of this study is to obtain infrared (IR) images and video and three-dimensional (3-D) scans of patients referred for biopsy based on the results of their diagnostic breast exam(s).

This research study is investigating infrared imaging (also referred to as infrared thermography, or digital infrared thermal imaging (DITI)) of breast cancer. The infrared images collected in this study will be used to construct a computational biothermal engineering model of the cancerous breast.

Patients will undergo standard breast cancer screening procedures as part of routine care at Parkland Comprehensive Breast Center. For any patients who are referred for biopsy based on the results of their breast cancer screening procedures, this research study will take infrared images of the patient. Patients will undergo infrared imaging prior to biopsy but will not delay biopsy or treatment; infrared images & video may be recorded at biopsy visit. The biopsy will confirm/diagnose whether the patient has a benign or malignant condition.

DETAILED DESCRIPTION:
The purpose of this research study is to obtain IR images, IR video, and 3-D scans of female patients' breasts (i.e., thermograms) who have been referred for biopsy based on the results of their diagnostic breast exams. These patients may be later diagnosed with a malignant or benign breast condition. The infrared images and video collected will be used to construct and validate a computational biothermal engineering model of breast cancer.

This research study does not involve any investigational drugs or treatments. This research study does not involve any FDA-approved drugs or devices.

In this research study, the equipment used (IR camera, 3-D scanner) will no be tested nor be used to diagnose or treat. Further, medical decisions will not be based on the use of these devices.

Infrared imaging (or digital thermal infrared imaging, DITI) is a non-invasive, non-contact, and harmless imaging procedure that measures the natural infrared radiation (body heat) emitted by the human body at normal 37°C body temperature. This procedure does not expose the patient to any radiation and is therefore entirely safe for the patient.

IR images and video will be obtained by IR equipment provided by University of Texas (UT) at Dallas researchers. IR equipment consists of an IR camera and ancillary equipment (e.g., tripod, computer, and vendor-provided IR image-processing software). The IR camera that will be used will be a commercial off-the-shelf product.

Additionally, a 3-D scanner will be used to obtain a 3-D surface contour map of the patient's breasts. This 3-D scanner is also non-invasive, non-contact, and does not expose the patient any radiation, similar to the IR camera. The 3-D scanner outputs a file format that is compatible with 3-D computer-aided design (CAD) software for engineering analysis.

ELIGIBILITY:
Inclusion Criteria:

* Females with a suspicious breast mass (BI-RADS 4C or 5).
* Referred for a breast biopsy.
* Capable of providing informed consent.

Exclusion Criteria:

* Currently undergoing treatment for breast cancer.
* Incapable of providing informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Spatial location of breast tumors | Two years
  Researchers will use subjects' radiological imaging data to quantify the location of the tumor inside the breast, including mammography, ultrasound, and/or magnetic resonance imaging (MRI), for patients who are diagnosed with breast cancer. The tumor location will be measured. The tumor location will serve as an input for the computational model. No diagnostic assessments will be made from these data for this research study.
3-D Surface contour maps of the breast | Two years
  Researchers will use a 3-D scanning device to reconstruct the 3-D surface geometry of subjects' breasts. The surface geometry of subjects' breasts will be measured. The surface geometry will serve as an input for the computational model. No diagnostic assessments will be made from these data for this research study.
Computational thermal model of breast cancer | Two years
  Researchers will use study data to validate a computational biothermal engineering model of the cancerous breast. The computational model will model and simulate the internal thermodynamic and heat transfer processes inside the breast with cancer. The model outputs expected surface temperatures of the breast with cancer. The model will be constructed using commercial engineering software, ANSYS Fluent. No diagnostic assessments will be made from these data for this research study.

CONTACTS AND LOCATIONS:
Overall Officials: Jody Hayes, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States